CLINICAL TRIAL: NCT02585375
Title: Latanoprost Preserved Versus Unpreserved: Effect on Tear Film Thickness as Measured With OCT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: OPHT-081214
Record Dates: First submitted 2015-04-26; First posted 2015-10-23 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with glaucoma or ocular hypertension 1 (Experimental): 35 patients with glaucoma or ocular hypertension
  Interventions: Drug: Preservative-free latanoprost 50µg/ml
- Patients with glaucoma or ocular hypertension 2 (Active Comparator): 35 patients with glaucoma or ocular hypertension
  Interventions: Drug: Preserved latanoprost 0.005%

INTERVENTIONS:
Drug: Preservative-free latanoprost 50µg/ml
  Arms: Patients with glaucoma or ocular hypertension 1
Drug: Preserved latanoprost 0.005%
  Arms: Patients with glaucoma or ocular hypertension 2

SUMMARY:
Topical antihypertensive eye drops are a key element of modern antiglaucoma treatment. Most of these eye drops contain preservatives to allow for the use of multi-dose containers. In the recent years evidence has, however, accumulated that these preservatives may induce ocular surface disease (OSD). This is particularly true for the most widely used preservative, benzalkonium chloride (BAK). Whereas this is well documented in many in vitro and animal studies, evidence from clinical trials is sparse. The only randomized masked study that showed superiority is a pivotal company-sponsored study indicating improved tolerability and reduced hyperemia of unpreserved versus preserved latanoprost eye drops.

The investigators have recently introduced an optical coherence tomography (OCT) technology that provides a resolution as high as 1.2 µm for the human cornea. Using this technology the investigators were able to show that tear film thickness (TFT) is negatively correlated with symptoms of OSD. Changes in TFT can be assessed with very high sensitivity below the level of resolution as also evident from studies after administration of lubricants.

In the present study, the investigators hypothesize that switching glaucoma patients from preserved prostaglandin analogues to unpreserved latanoprost is associated with an increase in TFT as measured with OCT. As a control the investigators will use preserved latanoprost and the study hypothesis will be tested in a randomized, controlled, single-masked parallel group design. TFT is chosen as main outcome variable, standard measures for signs and symptoms of OSD are selected as secondary outcomes. The present study may provide valuable information on the superiority of unpreserved versus preserved therapy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 years
* Diagnosed primary open angle glaucoma treated with preserved prostaglandin analogues containing at least 0.001% BAK for at least 6 months OR
* Patients with ocular hypertension treated with preserved prostaglandin analogues containing at least 0.001% BAK for at least 6 months
* IOP ≤ 21 mmHg in the study eye at the screening examination (under treatment)
* Mean tear film thickness at the screening visit < 4µm in the study eye

Exclusion Criteria:

* Participation in a clinical trial in the 3 weeks before the screening visit
* Severe visual field loss as defined as an MD of -15 or worse in the study eye
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Presence or history of a severe medical condition that will interfere with the study aim as judged by the clinical investigator
* Sjögren's syndrome
* Stevens-Johnson syndrome
* Presence or history of a severe ocular condition that will interfere with the study aim as judged by the clinical investigator
* Presence or history of allergic conjunctivitis
* Treatment with corticosteroids in the 4 weeks preceding the study
* Wearing of contact lenses
* Topical treatment with any ophthalmic drug in the 4 weeks preceding the study except glaucoma medication or topical lubricants
* Ocular infection
* Ocular surgery in the 6 months preceding the study (except laser trabeculoplasty)
* Pregnancy, planned pregnancy or lactating
* Contraindication against the use of topical prostaglandin therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-09-17 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09-02 (Estimated)

PRIMARY OUTCOMES:
Tear film thickness measured with high resolution optical coherence tomography (OCT) | 6 months

SECONDARY OUTCOMES:
Tear Break Up Time | 6 months
Tear Film Osmolarity | 6 months
Conjunctival hyperemia score | 6 months
Staining of the cornea with fluorescein according to Oxford scale | 6 months
Impression cytology according to Haller-Schober scale 2006 | 6 months
Schirmer 1 test | 6 months
Ocular Surface Disease Index score | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria